CLINICAL TRIAL: NCT04384679
Title: The Evaluation of Topical Hemostatic Powder Containing Hydrophilic Polymer With Potassium Ferrate for Hemostasis Following Nail Surgery
Brief Title: Benefit of Topical Hemostatic Powder Containing Hydrophilic Polymer With Potassium Ferrate for Hemostasis Following Nail Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to reallocation of resources, this study could not be initiated.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-02021562
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Nail Diseases
Keywords: Nails; Nail Surgery; Hemostasis; Potassium Ferrate
MeSH Terms: conditions — Nail Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Hydrophilic polymer and potassium ferrate powder (Experimental): Hydrophilic polymer with potassium ferrate powder is applied to the surgical wound with pressure until hemostasis is achieved
  Interventions: Device: Hydrophilic polymer and potassium ferrate powder
- Direct pressure with sterile gauze (No Intervention): Direct pressure with sterile gauze is applied to the surgical wound until hemostasis is achieved

INTERVENTIONS:
Device: Hydrophilic polymer and potassium ferrate powder — Application with pressure until hemostasis is achieved
  Arms: Hydrophilic polymer and potassium ferrate powder

SUMMARY:
The purpose of this study is to assess the efficacy and safety of topical hemostatic powder containing hydrophilic polymer with potassium ferrate for bleeding control after nail surgical procedures

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Patients scheduled for any type of nail surgical procedure
* Willingness to participate in the study
* Ability to understand all instructions in the English language

Exclusion Criteria:

* Failure to have nail surgery performed
* Likely inability to comply with the study protocol or cooperate fully with the research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Time (in seconds) to bleeding cessation with hydrophilic polymer and potassium ferrate; time (in seconds) to bleeding cessation with direct pressure with sterile gauze | Baseline
  Time (in seconds) will be measured from application of intervention/nonintervention until bleeding cessation

SECONDARY OUTCOMES:
Number of participants with at least one adverse event | End of study (28 days)
  Adverse events will only include those that are determined to be related to the study device

CONTACTS AND LOCATIONS:
Overall Officials: Shari R Lipner, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No